CLINICAL TRIAL: NCT02937064
Title: Multimodal Assessment of Knee Conditions
Acronym: MAKnee
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24302214
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Injury of Anterior Cruciate Ligament; Knee Injuries and Disorders
MeSH Terms: conditions — Osteoarthritis; Anterior Cruciate Ligament Injuries; Knee Injuries; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (6):
- Controls: Controls
- ACL subjects: Subjects with anterior cruciate ligament injuries.
- OA1, doubtful OA: Subjects with doubtful osteoarthritis.
- OA2, mild OA: Subjects with mild osteoarthritis.
- OA3, moderate OA: Subjects with moderate osteoarthritis.
- OA4, severe OA: Subjects with severe osteoarthritis.

SUMMARY:
The purpose of this study is to assess both osteoarthritis and other pathological knee conditions from the combination of signals that are known to provide information on the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 65

Exclusion Criteria:

* Rheumatoid arthritis
* Weight over 110 kg
* Previous total knee replacement surgery
* Contraindications to MRI

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls will be recruited using the newspaper advertisement. Subject with anterior cruciate ligament injuries will be recruited from the orthopaedic department and osteoarthritic subjects using patient Records of Oulu University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Severity of osteoarthritis (confirmed using X-ray and magnetic resonance imaging) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Simo Saarakkala, Ph.D., Principal Investigator — University of Oulu; Osmo Tervonen, M.D., Ph.D., Study Director — Oulu University Hospital
Locations (1):
- Univerisity of Oulu, Oulu, Finland